CLINICAL TRIAL: NCT06652828
Title: Training at the Limit of Balance Control on a Perturbation Treadmill to Prevent Unrecovered Falls in Geriatric Patients With and Without Cognitive Impairment
Brief Title: Perturbation-Based Treadmill Training to Prevent Unrecovered Falls in Geriatric Patients
Acronym: TRAIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oldenburg (Other)
Collaborators: Marienhospital Herne (Other); University of Ulm (Other); University of Konstanz (Other); University Hospital RWTH Aachen University, Aachen, Germany. (Unknown); Robert Bosch-Krankenhaus Stuttgart (Unknown); Heidelberg University Hospital, Heidelberg, Germany (Unknown); Technische Hochschule Ulm (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. med. Tania Zieschang, Prof. Dr. med., University of Oldenburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-UOL-MG-005-01; 01KG2303 (Other Grant/Funding Number: BMBF)
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Fall Prevention; Exercise; Geriatrics; Cognitive Impairment; Perturbation
Keywords: treadmill; unrecovered falls; fall risk; training; falls; balance; rehabilitaion
MeSH Terms: conditions — Motor Activity; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Treadmill Training (CTT) (Active Comparator)
  Interventions: Other: Conventional Treadmill Walking (CTT)
- Perturbation-Based Balance Training (PBT) (Experimental)
  Interventions: Other: Perturbation-Based Balance Training (PBT)

INTERVENTIONS:
Other: Conventional Treadmill Walking (CTT) — The CTT serves as a comparison to PBT. It involves standard treadmill walking without perturbations on the same treadmill. This intervention is conducted over the same defined period as PBT (3-6 weeks), with a matched frequency and exercise time compared to the PBT group for consistency. Participants are secured with safety harnesses while walking.
  Other Names: Exercise intervention
  Arms: Conventional Treadmill Training (CTT)
Other: Perturbation-Based Balance Training (PBT) — Overall, 9 training sessions with different objectives and progression regarding perturbation directions, predictability, and intensity will be conducted within 3-6 weeks. During the initial sessions, familiarizing participants with the treadmill and establishing their individual walking pace will be focused. Pace can be individually adjusted in each training session. Participants are secured with safety harnesses while walking.
  Other Names: Gait adaptability training; Reactive balance training
  Arms: Perturbation-Based Balance Training (PBT)

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of perturbation-based balance training (PBT) in preventing unrecovered falls among geriatric patients aged ≥70 years with a prospective fall risk of ≥40%. The study will also assess the safety and feasibility of PBT. The main research questions are:

A total of 396 participants will receive 9 training sessions of either PBT or conventional treadmill training and will attend an assessment before and after the intervention, as well as 6 and 12 months follow up. Falls will be documented throughout the entire study period using calendars, telephone interviews, and proxy information. The primary outcome, unrecovered falls, will be recorded after the end of the intervention until 12 months follow up.

DETAILED DESCRIPTION:
Falls are common and the leading cause of injuries among older adults, but falls may be attenuated by the promising and time-efficient intervention called perturbation-based balance training (PBT). The aim of the TRAIL-study is to confirm the effectiveness of a treadmill PBT protocol for preventing unrecovered falls in geriatric patients with and without cognitive impairment. This study is designed as a confirmatory, multicenter, assessor-blinded, randomized controlled study. The 396 geriatric patients aged ≥70 years with ≥40% prospective fall risk and being capable of walking ≥70 m in a 2-Minute Walk Test will receive 9 sessions of PBT on a treadmill (intervention) or a conventional treadmill training (control group; CTT).

Outcome assessments will be performed shortly after the intervention interval as well as 6 and 12 months thereafter. The primary outcome is defined as unrecovered falls (defined as falls in which persons who fell are unable to get up independently) within 12-month follow-up. Falls are documented over at least 12 months using calendars, telephone interviews, and proxy information. Secondary outcomes include mobility, balance performance, concerns about falling, physical activity and capacity, stepping responses, health-related quality of life, cognitive functioning, mobility, reactive dynamic balance and training acceptability of PBT. The study will be accompanied by a patient advisory board and an expert advisory board and focus groups will be conducted to involve the target group.

Based on pilot studies and the available literature, we expect a ≥50% reduction of unrecovered falls during the following year in the intervention group (PBT) compared to the control group (CTT).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 70 years
* ≥40% prospective fall risk for the following year according to the Fall Risk Assessment Tool (FRAT-up)
* Walking distance ≥ 70 m in the 2 Minute Walk Test
* Possibility to reach the study site at least via taxi
* Written informed consent, obtained according to international guidelines and local laws

Exclusion Criteria:

* MoCA score < 10 pts (or MMSE < 17 pts)
* Performing a Timed up and Go test (TUG) <10 s
* Leg amputation
* Osteosynthesis or joint replacement of lower extremities within the past 6 weeks.
* Blindness
* Parkinson's disease with Hoehn and Yahr stage > 3
* Body weight >135 kg and height >185 cm
* Life-expectancy <12 months, instable or severe illness
* Inability to communicate verbally and coorporate appropriatly
* (Prior) participation perturbation training programs
* Gait-relevant foot-drop paresis

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of unrecovered falls | Continuously from intervention end until 12 months after the end of the intervention
  Falls are assessed using fall calendars, telephone interviews, and proxy information.

SECONDARY OUTCOMES:
Rate of falls | Continuously from intervention end until 12 months after the end of the intervention
  Falls are assessed using fall calenders, telephone interviews, and proxy information.
Physical activity | Before the training intervention (up to 4 weeks before the beginning of the training), after the intervention (up to 8 weeks after its beginning), 6 months after the intervention, and 12 months after the intervention
  Physical activity will be measured over 7 days using a body-fixed inertial measurement unit (AX6, Axivity Ltd., Newcastle, UK) , which will be placed at lumbar level (L5) of the participant. The sensor measures linear acceleration data in 3 dimensions in combination with angular data. From these data, besides others, time spent with physical activity, steps as well as time spent in the supine sitting or standing position can be determined and reported. Data will be used to describe the participants and to report falls per physical activity.
Stepping response (a) | 12 months after the intervention
  Modified Stepping Threshold Tests (i.e. single step, multiple step threshold). Participants will experience suface perturbations in ante-posterior as well as mediolateral direction with increasing intensity until they have to perform a single compensatory step or multiple steps to recover balance. Higher perturbation levels for the single or multiple step threshold indicate better static reactive balance.
Stepping reponse (b) | Before the training intervention (up to 4 weeks before the beginning of the training), after the intervention (up to 8 weeks after its beginning), 6 months after the intervention, and 12 months after the intervention
  Choice Stepping Reaction Test
Cognitive functioning (a) | Before the training intervention (up to 4 weeks before the beginning of the training), and 12 months after the intervention
  Montreal Cognitive Assessment (MoCA). Minimum value: 0 points; Maximum value: 30 points; higher values indicate better cognitive functioning.
Cognitive functioning (b) | Before the training intervention (up to 4 weeks before the beginning of the training), after the intervention (up to 8 weeks after its beginning), 6 months after the intervention, and 12 months after the intervention
  TMT (Trail Making Test)
Concerns about falling | Before the training intervention (up to 4 weeks before the beginning of the training), after the intervention (up to 8 weeks after its beginning), 6 months after the intervention, and 12 months after the intervention
  Short Falls Efficacy Scale International (Short FES-I). Minimum value: 7 points, Maximum value: 28 points; higher values indicate more concerns about falling.
Health-related quality of life | Before the training intervention (up to 4 weeks before the beginning of the training), after the intervention (up to 8 weeks after its beginning), 6 months after the intervention, and 12 months after the intervention
  Euro Quality of Life with visual analogue scales (EQ-VAS), values of 0-100: lower values indicate worse subjective health; EuroQol 5-Dimensions 5-Levels
Physical capacity (a) | Before the training intervention (up to 4 weeks before the beginning of the training), after the intervention (up to 8 weeks after its beginning), 6 months after the intervention, and 12 months after the intervention
  2MWT (2 Minute Walk Test )
Physical capacity (b) | Before the training intervention (up to 4 weeks before the beginning of the training), after the intervention (up to 8 weeks after its beginning), 6 months after the intervention, and 12 months after the intervention
  SPPB (Short Physical Performance Battery), including balance, leg strength and gait speed; minimum value: 0 points; maximum value: 12 points; higher values indicate better physical capacity.
Physical capacity (c) | Before the training intervention (up to 4 weeks before the beginning of the training), after the intervention (up to 8 weeks after its beginning), 6 months after the intervention, and 12 months after the intervention
  TUG (Timed "Up and Go"-Test)
Nutritional status | Before the training intervention (up to 4 weeks before the beginning of the training), 6 months after the intervention, and 12 months after the intervention
  MNA (Mini Nutritional Assessment); values of 0-30: lower values indicate worse nutritional status
Reactive dynamic balance (a) | 3rd (during the on average 1st week of the intervention) and last training session (during the on average 3rd week, at maximum 6th week of the intervention) (intervention group only), and 12 months after the intervention (intervention and control group)
  Adapted Compensatory Arm and Leg Movements after perturbations induced on the treadmill during walking. Minimum value: 16 points; Maximum value: 108 points; higher values indicate better reactive dynamic balance.
Reactive dynamic balance (b) | 3rd (during the on average 1st week of the intervention) and last training session (during the on average 3rd week, at maximum 6th week of the intervention) (intervention group only), and 12 months after the intervention (intervention and control group)
  Spatio-temporal, kinematic and stability parameters (video-based, inertial measurement units and center of pressure data)
Laboratory falls | during 3rd (on average 1st week of the intervention) and last training session (on average 3rd week, at maximum 6th week of the intervention; intervention group only), and 12 months after the intervention (intervention and control group)
  Falls after perturbations on the treadmill. A fall is determined based on video recordings. A fall is defined as unambiguous support by the safety harness after the perturbation.
Acceptability of PBT | during the last training session (during the on average 3rd week, at maximum 6th week of the intervention, in the intervention group only)
  Theoretical Framework of Acceptability-based Questionnaire
Vibration sensation | Before the training intervention (up to 4 weeks before the beginning of the training), after the intervention (up to 8 weeks after its beginning), 6 months after the intervention, and 12 months after the intervention
  Vibration measurement at the inner ankle using a tuning fork. Minimum value: 1 point, Maximum value: 8 points; higher values indicate higher sensation

OTHER OUTCOMES:
Assessment of safety | Continuously from baseline assessment until 12 months after the end of the intervention (intervention starts at maximum 4 weeks after baseline assessment)
  Intervention-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tania Zieschang, Prof. Dr. med., Principal Investigator — Carl von Ossietzky University Oldenburg
Locations (3):
- Germany (3):
  - Geriatric Center, Heidelberg University Hospital, Agaplesion Bethanien Krankenhaus, Heidelberg, Baden-Wurttemberg
  - Department of Geriatric Medicine, University Hospital Marien Hospital Herne - Ruhr-University Bochum, Herne, North Rhine-Westphalia
  - Carl von Ossietzky Universität, Department für Versorgungsforschung, Abteilung Geriatrie, Oldenburg

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request via e-mail.
Supporting Information: Study Protocol
Time Frame: The data will be available for 10 years after the last publication of the study results.
Access Criteria: Data will be made available upon reasonable request via e-mail.

REFERENCES:
- [Derived] Koschate-Storm J, Werner C, Bartel J, Bauer JM, Becker C, Drefs S, El-Seoud N, Giehl C, Hackbarth M, Hezel N, Klenk J, Trampisch U, Wirth R, Zieschang T, Schwenk M. Treadmill perturbation-based balance training to prevent unrecovered falls in fall-prone older adults with and without cognitive impairment: protocol for the multi-center randomized controlled TRAIL study. BMC Geriatr. 2025 Dec 23. doi: 10.1186/s12877-025-06599-w. Online ahead of print. PMID 41436967
- See also: Related Info — https://uol.de/geriatrie/projekte/trail